CLINICAL TRIAL: NCT01500005
Title: The Effect of Vitamin D Supplementation on Arterial Stiffness, Blood Pressure, Oxidative Stress and Inflammation in Diabetic Patients
Brief Title: The Effect of Vitamin D Supplementation on Arterial Stiffness in Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Fany Tusia, medical center, Assaf-Harofeh Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: shlomit10
Record Dates: First submitted 2010-12-15; First posted 2011-12-26 (Estimated); Last update posted 2011-12-26 (Estimated); Status verified 2011-12

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- vitamin D (Experimental): Baby D3 drops
  Interventions: Drug: Baby D3 drops

INTERVENTIONS:
Drug: Baby D3 drops — 2000-4000 iu per day
  Other Names: vitamin D

SUMMARY:
The incidence of type 2 Diabetes Mellitus is increasing at an alarming rate worldwide.

Cardiovascular disease is the leading cause of death in patients with type 2 diabetes.

Recently, increasing amount of evidence suggests that vitamin D may influence various nonskeletal medical conditions, including cardiovascular disease, hypertension, diabetes, cancer, autoimmune disorders and more. The purpose of this trial is to investigate the effect of vitamin D supplementation on 24 hours blood pressure monitoring, arterial stiffness, oxidative stress and inflammation in vitamin D deficient diabetic patients.

DETAILED DESCRIPTION:
Background:

The incidence of type 2 Diabetes Mellitus is increasing at an alarming rate worldwide, with more than 1 million new cases per year diagnosed in the United States alone. [1] Diabetes is the fifth leading cause of death in the United States, and it is also a major cause of significant morbidity.

Cardiovascular disease is the leading cause of death in patients with type 2 diabetes.

The risk of Cardiovascular disease (CVD) mortality in type 2 diabetic patients is more than double compared with that in age-matched subjects. [2] Therefore, reducing cardiovascular risk in diabetic patients is of great importance.

Vitamin D3 (cholecalciferol), the most powerful form of vitamin D, is synthesized in the skin from 7-dehydrocholesterol by action of sunlight (ultraviolet B radiation). Vitamin D3 is biologically inert. In the hepatic parenchyma, vitamin D3 is converted to 25-hydroxyvitamin D3 (25OHD3) and must be converted to the active hormone 1,25-dihydroxy vitamin D (calcitriol). 25OHD is the most plentiful and stable metabolite of vitamin D. As such, the 25OHD level in the serum is the best indicator of vitamin D level. [3]

The major and most well known function of Vitamin D is to maintain calcium and phosphorus homeostasis and promote bone mineralization. It is well understood that vitamin D deficiency leads to osteomalacia and osteoporosis in adults. [4]

However, recently, increasing amount of evidence suggests that vitamin D may also influence various nonskeletal medical conditions, including cardiovascular disease, hypertension, diabetes, cancer, autoimmune disorders and more [4, 5] An evolving data indicates that vitamin D deficiency is much more prevalent than previously recognized. In the United States, as well as in other parts of the world, the mean population serum 25OHD levels have decreased in the last decade. The best example of this drop comes from the National Health and Nutrition Examination Survey (NHANES) population showing near doubling in the number of subjects in the American population from 1994 to 2004 with 25OHD levels less than 30 ng/ml.[6]

The possible explanations for this dramatic decrease in vitamin D level are: downward in milk consumption, upward in sun protection and upward in obesity. [7]

All cause and cardiovascular mortality:

The NHANES III database clearly shows an increase in adjusted all cause mortality as the serum 25OHD level falls to less than 30 ng/ml, especially in woman, and peak protection from death with a 25OHD level in the 35-40 ng/ml range. The prevalence of coronary artery disease, heart failure, and peripheral artery disease is significantly increased in a stepwise fashion as the serum 25OHD level drops to less than 30 and then 20 ng/ml (insufficiency and deficiency, respectively). [8]

A recent meta-analysis of 18 trials comprising 57,311 randomly assigned participants, found that vitamin D supplementation >500 IU/day reduced all cause mortality by 7%, in part by decreasing CV deaths.[9] Deficient or insufficient serum 25(OH) D levels have been documented in patients with myocardial infarction .[10] A correlation between vitamin D deficiency and subsequent major adverse CV events was found among the 1739 Framingham Offspring Study participants who were free of CV disease at baseline. In this prospective observational study, 25(OH) D levels were measured at baseline and subjects were followed up for a mean of 5.4 years. The rate of a composite CV end point (fatal or nonfatal MI, ischemia, stroke, or heart failure) was 53% to 80% higher in people with low vitamin D levels.[11]

The reason for this association between all cause mortality, CVD and vitamin D insufficiency/deficiency is unclear. It is also unclear whether vitamin D supplementation will normalize the CVD risk in these patients.

In a recent systemic review Wang et al found no completed trials that have tested the effect of vitamin D and calcium supplementation on CVD as the primary end point. [12]

Vitamin D and diabetes Inspection of the recent vitamin D insufficiency/deficiency epidemiological literature has brought to light the striking inverse correlation of the25OHDlevel not only to cardiovascular disease but also to essentially all of the elements of the human metabolic syndrome: hypertension; obesity; insulin resistance and glucose Intolerance [3] Likewise, in cross sectional studies, inverse associations between serum 25(OH) D and presence of type 2 diabetes have been reported in a variety of cohorts. [13-15]

One example is the analysis of data from participants who attended the morning examination of the Third National Health and Nutrition Examination Survey (1988-1994) that showed an inverse association between vitamin D status and diabetes.[13]

This observations regarding the high prevalence of vitamin D deficiency among type 2 DM patients do not establish causative relationship between the two.

In the women's Health Study, an intake of 511 IU/d of vitamin D or more was associated with lower risk of incidence type 2 DM compared with low intake [16]

Vitamin D and Arterial stiffness Augmentation pressure, reflecting the pulsatile component of blood pressure and thus arterial stiffness, is a well-known risk factor for cardiovascular disease and outcome.[17-21] Augmentation index (AIx), a non invasive measure of arterial stiffness, has been shown to predict coronary artery disease (CAD) in the general population and in patients with type 2 diabetes [20, 22, 23] The differential effects on arterial stiffness may be responsible for the different impact of diverse antihypertensive drug/treatments on CAD.[21] Different drugs have been proved to improve arterial stiffness. One example is the beneficial effect of statins on AIx, a result that is independent of their cholesterol lowering effect. [24] Andrade et al found that Lower 1,25-OH2D3 levels were associated with higher Aix in 131 outpatients identified from individual cardiac or kidney disease clinics. [25] Vitamin D regulates the renin-angiotensin system (RAS) in experimental animals. Recently data in humans suggest that low plasma 25-hydroxyvitamin D levels may result in upregulation of the RAS in otherwise healthy humans. [26] No studies to date examined the effect of vitamin D supplementation on blood pressure and arterial stiffness as primary end point.

The purpose of this trial is to investigate the effect of vitamin D supplementation on 24 hours blood pressure monitoring, arterial stiffness, oxidative stress and inflammation in vitamin D deficient diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients
* Aged 18 years or older
* VITAMIN d deficiency

Exclusion Criteria:

* CCT<30
* A history of treatment with vitamin D supplementation in the last 3 months
* Treatment with nitrates
* Uncontrolled heart failure
* Uncontrolled hypertension and/or any change in the hypertensive medications during the last 1 month.
* Any malignancy with life expectancy of less then 1 year
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2010-08; Primary Completion 2011-01 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
arterial stiffness | 3 months

SECONDARY OUTCOMES:
blood pressure holter | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Shlomit koren, MD, Principal Investigator — Department of Internal Medicine A , Research & Development unit Assaf Harofeh Medical Center, Zerifin, affiliated to Sackler School of Medicine, Tel Aviv, Israel
Locations (1):
- Department of Internal Medicine A , Research & Development unit Assaf Harofeh Medical Center, Zerifin, affiliated to Sackler School of Medicine, Tel Aviv, Israel, Ẕerifin, Zerifin, Israel